CLINICAL TRIAL: NCT03129477
Title: TELE-monitoring in Chronic Obstructive Pulmonary Disease
Acronym: TELECOPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Conde, Bebiana, M.D. (Individual)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2016-03-26; First posted 2017-04-26 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: COPD
Keywords: Non invasive ventilation in COPD; Noninvasive ventilation; Tele-monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Computorizada randomizados selection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring in NonInvasiveVentilation (Experimental): Tele-monitoring in noninvasive ventilation with Lumis 150 and others Resmed equipments with AirView monitoring system, in COPD patients.
  • Education and adaptation of the patient to NIV.
  Interventions: Procedure: Telemonitoring in noninvasive ventilation
- 2- conventional monitoring group (No Intervention): Conventional monitoring group
  • Education and adaptation of the patient to NIV.

INTERVENTIONS:
Procedure: Telemonitoring in noninvasive ventilation — Compare telemonitoring to conventional monitoring to optimize Ventilation
  Arms: Telemonitoring in NonInvasiveVentilation

SUMMARY:
COPD is the fourth cause of death worldwide and it is expected to be the third in 2020.

Non-invasive ventilation (NIV) has a positive impact in reducing mortality related to chronic respiratory failure in stable patients with COPD. Moreover, the addition of home NIV to home oxygen therapy reduces hospital admissions and improves patients outcomes.

Patients monitoring is crucial. It is increasingly recognized the potential of telemedicine in reducing morbidity and mortality, as well as healthcare utilisation and its associated costs. In particular, home telemonitoring (TM)- a technology measuring patients'clinical parameters and symptoms at home and allowing communication between healthcare professionals and patients over distance- has gained much attention. However, despite a growing body of evidence for TM in the management of COPD and other chronic diseases, the benefit of telemonitoring for Home mechanical ventilation concerning clinical and economic outcomes remains to be clearly demonstrated.

The study aims to assess the impact that telemonitoring would have NIV efficacy, patient quality of life and satisfaction, through a prospective randomized study.The primary endpoint is the time for appropriate adaptation and therapy efficacy, defined as average SatO2 to 90% in 24h oximetry.

DETAILED DESCRIPTION:
A prospective randomized study, with 2 branches.

The primary endpoint is the time for appropriate adaptation and therapy efficacy, defined as average SatO2 to 90% in 24h oximetry.

Patients with COPD (n=100) based in Gold 2017. Patients with stable COPD and Pa CO2 > 52 mmHg in blood gases. These patients might have a polygraph or polysomnographic sleep study AHI/RDI < 15/h

1. 1st hospital visit - D0- Inclusion criteria Confirmation; Randomization to 2 groups (1 - telemonitoring group (TM group) with the equipment Lumis 150, Stellar 150 or ventilator Astral 150 with AirView system; 2 - conventional monitoring group (CM group); Mode and settings titration will be selected according to patients needs and tolerance; Education and adaptation of the patient to VNI and optimize ventilation.
2. 2nd home healthcare professionals visit (D 1M)-
3. 3th hospital visit- D 3M- Compliance and ventilation effectiveness assessment (24 oximetry and ventilator data analysis); Settings adjustment if required;
4. 4th hospital visit - D 6M- Compliance and ventilation effectiveness assessment (24 oximetry and ventilator data analysis) ; Settings adjustment if required
5. 5th hospital visit - D 12M- Compliance and ventilation effectiveness assessment (24 oximetry and ventilator data analysis); Settings adjustment if required

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD (n=100) based in Gold 2017. Patients with Stable COPD and PaCO2 > 52 mmHg in blood gases. These patients might have a polygraph or polysomnographic sleep study AHI/RDI <15/h

Exclusion Criteria:

* Patients with ventilatory treatment;
* Without diagnosis of COPD
* Polygraph or polysomnographic sleep study AHI/RDI >=15/h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Time for appropriate adaptation and therapy efficacy | one year
  Calculate the time required to achieve a 4-hour-day adherence on 70% of the days and a sato2 <90% in less than 10% of the time in 24-hour oximetry.

SECONDARY OUTCOMES:
Rate of readmissions for COPD acute exacerbations and mortality | One year
  Calculate the hospital readmission rate by COPD acute exacerbations and mortality for 1 year and compare these rates between the 2 intervention groups (conventional monitoring and telemonitoring)

CONTACTS AND LOCATIONS:
Overall Officials: Bebiana Conde, MD, Principal Investigator — Centro Hospitalar Tras-os-Montes e Alto Douro
Locations (1):
- Centro Hospitalar Tras-os-Montes e Alto Douro, Vila Real, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Clinical data of the patients are required to adjust the ventilation parameters.

REFERENCES:
- [Background] Kohnlein T, Windisch W, Kohler D, Drabik A, Geiseler J, Hartl S, Karg O, Laier-Groeneveld G, Nava S, Schonhofer B, Schucher B, Wegscheider K, Criee CP, Welte T. Non-invasive positive pressure ventilation for the treatment of severe stable chronic obstructive pulmonary disease: a prospective, multicentre, randomised, controlled clinical trial. Lancet Respir Med. 2014 Sep;2(9):698-705. doi: 10.1016/S2213-2600(14)70153-5. Epub 2014 Jul 24. PMID 25066329
- [Background] Struik FM, Sprooten RT, Kerstjens HA, Bladder G, Zijnen M, Asin J, Cobben NA, Vonk JM, Wijkstra PJ. Nocturnal non-invasive ventilation in COPD patients with prolonged hypercapnia after ventilatory support for acute respiratory failure: a randomised, controlled, parallel-group study. Thorax. 2014 Sep;69(9):826-34. doi: 10.1136/thoraxjnl-2014-205126. Epub 2014 Apr 29. PMID 24781217
- [Background] McEvoy RD, Pierce RJ, Hillman D, Esterman A, Ellis EE, Catcheside PG, O'Donoghue FJ, Barnes DJ, Grunstein RR; Australian trial of non-invasive Ventilation in Chronic Airflow Limitation (AVCAL) Study Group. Nocturnal non-invasive nasal ventilation in stable hypercapnic COPD: a randomised controlled trial. Thorax. 2009 Jul;64(7):561-6. doi: 10.1136/thx.2008.108274. Epub 2009 Feb 12. PMID 19213769